CLINICAL TRIAL: NCT03054818
Title: Safety Evaluation of China Patients: Long-term Treatment Outcome of Conbercept Ophthalmic Injection in Real Word
Brief Title: Safety Evaluation of China Patients: Long-term Treatment Outcome of Conbercept Ophthalmic Injection in Real Word（STONE）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RG01N-1578-1.0
Record Dates: First submitted 2017-02-08; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Wet Age-related Macular Degeneration (wAMD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a post-marketing drug safety monitoring study in a prospective manner, and data collection will be performed in a registration-follow-up manner. Safety information about patients who have received intravitreal injection of Conbercept Ophthalmic Injection in medical institutions involved in the study during research will be actively monitored without intervening in diagnosis and treatment. All patients enrolled will be followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

1. The condition that informed consent has been freely given prior to research-related procedures;
2. Patients who have received at least one intravitreal injection of Conbercept Ophthalmic Injection after informed consent has been given.

Exclusion Criteria:

1. Patients who have been on any of other anti-VEGF drugs systematically or locally, including but not limited to bevacizumab, ranibizumab and aflibercept, 90 days before enrollment;
2. Those who are on other study drugs or have been on other study drugs 30 before informed consent is given.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All medical academies will initially identify whether patients are enrolled based on baseline registration information.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
New Adverse Reactions | 1 year
  To observe the type, incidence and severity of new adverse reactions in patients who have received intravitreal injection of Conbercept Ophthalmic Injection during the study;
Common Ocular Adverse Events | 1 year
  To observe the type, incidence and severity of common ocular adverse events in patients who have received intravitreal injection of Conbercept Ophthalmic Injection during the study, including: 1) bleeding at injection site; 2) increased intraocular pressure (IOP); 3) conjunctival congestion; 4) conjunctivitis; 5) decreased visual sensitivity; and 6) muscae volitantes.
Common Ocular Adverse Events | 1 year
  To evaluate the Common Ocular AEs' correlation with Conbercept Ophthalmic Injection therapy.

SECONDARY OUTCOMES:
Other Ocular Adverse Events | 1 year
  To observe the type, incidence and severity of other ocular adverse events in patients who have received intravitreal injection of Conbercept Ophthalmic Injection during the study.
Other Ocular Adverse Events | 1 year
  To evaluate the Other Ocular AEs' correlation with Conbercept Ophthalmic Injection therapy.
Non-ocular Adverse Events | 1 year
  To observe the type, incidence and severity of non-ocular adverse events during the study
Non-ocular Adverse Events | 1 year
  To evaluate the Non-ocular AEs' correlation with Conbercept Ophthalmic Injection therapy.
Adverse Events of Special Interest(AESI) | 1 year
  To observe the incidence and severity of adverse events of special interest (AESI) during the study, including: 1) retinal detachment; 2) retinal tears; 3) retinal pigment epithelial detachment; 4) retinal pigment epithelium tears; 5) geographic atrophy; 6) endophthalmitis; 7) arterial thromboembolic events (ATEs); and 8) hypertension
Adverse Events of Special Interest(AESI) | 1 year
  To evaluate the AESI's correlation with Conbercept Ophthalmic Injection therapy.
SAE | 1 year
  To observe the type, incidence and severity of all severe adverse events during the study
SAE | 1 year
  To evaluate the SAEs' correlation with Conbercept Ophthalmic Injection therapy.
Adverse Events Related to Intravitreal Injection Practices | 1 year
  To observe the incidence and severity of possible adverse events related to intravitreal injection practices of Conbercept Ophthalmic Injection during the study.
Adverse Events of Special Population | 1 year
  To observe the incidence and severity of adverse events of special population during the study,including children and adolescents (aged under 18), and pregnant women.
Adverse Events of Special Population | 1 year
  To evaluate the AEs' correlation with Conbercept Ophthalmic Injection therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ningli Wang, Principal Investigator — BEIJING TONGREN HOSPITAL, CMU
Locations (49):
- China (49):
  - Baoji People'S Hospital, Baoji
  - Beijing Aier-Intech Eye Hospital, Beijing
  - Beijing Tongren Hospital, Cmu, Beijing
  - Eye Hospital, China Academy of Chinese Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The 306Th Hospital of Pla, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The third people's Hospital of Dalian, Dalian
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Second Affiliated Hospital of ZhejiangUniversity School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - JOINT SHANTOU INTERNATIONAL EYE CENTER of Shantou University and The Chinese University of Hong Kong, Hong Kong
  - Shandong Eye Hospital, Jilancun
  - Shandong Provincal Hospital, Jilancun
  - The Second Hospital of Jilin University, Jiling
  - Kashgar First People's Hospital, Kashgar
  - Lanzhou University Second Hospital, Lanzhou
  - Central Hospital of Mudanjiang Forestry, Mudanjiang
  - Jiangsu Province Hospital of CTM, Nanjing
  - The People'S Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Ningbo Eye Hospital, Ningbo
  - Ningxia People'S Hospital, Ningxia
  - Pingdingshan People'S Hospital No.1, Pingdingshan
  - The First Hospital of Qiqihar, Qiqihar
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Baoshan Hospital of Integrate Traditional Chinese and Western Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Tongji Hospital, Shanghai
  - Shenyang the Fourth Hospital of People, Shenyang
  - The Fourth Affiliated Hospital of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Shenzhen Eye Hospital, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Eye Hospital, Taiyuan
  - Tianjin Medical University Eye Hospital, Tianjin
  - No.474 Hospital of Pla, Ürümqi
  - Wuhan General Hospital of Pla, Wuhan
  - Wuxi NO.2 People's Hospital, Wuxi
  - Tangdu Hospital, Xi'an
  - Xi'An No.4 Hospitla, Xi'an
  - Xijing Hospital, Xi'an
  - Hebeisheng Eye Hospital, Xingtai
  - The First People's Hospital of Xuzhou, Xuzhou
  - Zhongshan Ophthalmic Center, Sun Yay-Sen University, Zhongshan

IPD SHARING:
Plan to Share IPD: Undecided